CLINICAL TRIAL: NCT02066155
Title: Ongoing Diabetes Self-Management Support in Church-Based Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Gretchen Piatt, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-PAF00455 PAF; DSMS (Other Grant/Funding Number: Bristol-Myers Squibb Foundation)
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes
Keywords: diabetes self-management support; diabetes-related distress; parish nurses; peer support
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Parish nurse (Experimental): On-going support provided by parish nurse
  Interventions: Behavioral: Parish nurse
- Peer support (Experimental): On-going support provided by a person with diabetes
  Interventions: Behavioral: Peer Support
- Control group (No Intervention): No on-going support provided

INTERVENTIONS:
Behavioral: Parish nurse — On-going support following diabetes self-management education provided by Parish Nurse
  Arms: Parish nurse
Behavioral: Peer Support — On-going support following diabetes self-management education provided by a trained person with diabetes
  Arms: Peer support

SUMMARY:
African Americans are twice as likely to have diabetes compared to their White counterparts and experience higher rates of diabetes-related complications. Diabetes-related health disparities underscore the need for effective, culturally tailored approaches to promote and sustain diabetes self-management over time. Diabetes self-management education (DSME) is effective in improving diabetes outcomes in the short-term. However, many adults with diabetes cannot sustain achieved improvements without continued follow-up and support. The 2012 revisions of both the National Standards for Diabetes Care 6 and the National Standards for DSME and Support emphasize the importance of providing both initial DSME and on-going diabetes self-management support (DSMS) to assist people with diabetes in maintaining effective self-management throughout a lifetime. While a great deal is understood about how to provide effective, initial DSME, less is known about who, where, when, and how to provide effective, sustained DSMS. One significant challenge is that DSME is a covered benefit in the healthcare system, while DSMS is not. This ultimately limits access and availability of DSMS programs, especially for low-income African Americans. Accordingly, there is critical need to develop, evaluate, and understand effective DSMS models that are ongoing, patient-driven, and embedded in the community.

DETAILED DESCRIPTION:
The long-term goal of our research is to determine the most effective, practical, and sustainable approaches to provide ongoing DSMS in the context of the communities in which people live. In the African American community, the church plays a central role in community life and can serve as a powerful channel to deliver health promotion programs. Churches in the community are thus ideal venues to intervene to help people with diabetes achieve their self-management related goals. The objective of this proposal is to examine the relative effectiveness of three approaches to address DSMS compared to enhanced usual care within the context of the church-based setting. To accomplish this objective, a cluster randomized, modified stepped wedge, practical behavioral trial with three parallel DSMS approaches will be implemented. Twenty-one African American churches (23 African American participants per church) in metro-Detroit will be randomized to one of three DSMS approaches. Fourteen parish nurses who are volunteers at the churches, and 21 peer leaders will be trained to deliver DSMS. Measures will be collected at baseline, 6, 9, 15 and 27-month follow-up. The primary outcome will be changes in A1c at 9, 15 and 27-month follow-up. Secondary outcomes include changes in weight, blood pressure, quality of life, and diabetes related distress at 9,15 and 27-month follow-up. We hypothesize that 1) participants in both Parish Nurse DSMS and Peer Leader DSMS will have improved outcomes over enhanced usual care, and that 2) participants in Parish Nurse + Peer Leader DSMS will sustain improvements in outcomes achieved following DSME at significantly higher levels than participants in Parish Nurse DSMS and Peer Leader DSMS

ELIGIBILITY:
Inclusion Criteria for Parish Nurses

* Registered nurse in Michigan
* Identified as a parish nurse in the participating church
* Member of the Detroit Parish Nurse Network
* Willing to serve as a parish nurse for the research study

Inclusion Criteria for Peer Leaders

* Have diabetes ≥ one year
* Be a resident of metro-Detroit

  -≥21 years old and ≥ 8th grade education
* Have transportation to attend training
* Be willing to commit to 3 months of training
* Actively working on his/her own self management goals and
* Willing to serve as a peer leader

Inclusion Criteria for Participants

* Have diabetes ≥ 6 months
* Resident of metro-Detroit

  -≥ 21years old
* Be under the care of a physician for diabetes
* Have transportation to attend the program
* Be a member or regularly attend the participating church

Exclusion Criteria for Parish Nurses

* Not a registered nurse
* Not a parish nurse in the church
* Not a member of the DPNN
* Unwilling to serve as a parish nurse for the research studyExclusion Criteria for Participants:
* Non ambulatory or serious health conditions or psychiatric illness (severity requiring hospitalization)
* Serious diabetes complications (e.g. blindness) that would impede meaningful participation

Exclusion Criteria for Peer Leaders and Participants:

* Non ambulatory or serious health conditions or psychiatric illness (severity requiring hospitalization)
* Serious diabetes complications (e.g. blindness) that would impede meaningful participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | Baseline, 3, 9, 15, 27 months
  Measure of long-term glucose control

SECONDARY OUTCOMES:
BMI | Baseline, 3, 9, 15, 27 months
  Measure of weight loss

OTHER OUTCOMES:
Diabetes-related distress | Baseline, 3, 9, 15, 27 months
  Measure of psychological distress caused by diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen A Piatt, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical School, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No